CLINICAL TRIAL: NCT00730704
Title: Acceptance of Human Papillomavirus Vaccination in Postpartum Women
Acronym: HPV Acceptance
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jason D. Wright, Assistant Professor of Gynecologic Oncology, Columbia University
Other Study IDs: AAAD1877
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Human Papilloma Virus; HPV; Post Partum
Keywords: Human Papilloma Virus vaccines; HPV; Gardasil; Post partum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Worldwide cervical cancer remains a major cause mortality among women. It is estimated that each year over 490,000 women are diagnosed with cervical cancer and more than 270,000 die from the disease. While the implementation of widespread screening programs has reduced the burden of cervical cancer, a large percentage of the population still remains unscreened or is underscreened. It is now recognized that human papillomavirus (HPV) is a necessary precursor for the development of cervical cancer. The first vaccine to prevent HPV was recently approved by the Food and Drug Administration and is now available at doctors offices. Despite the availability of a safe and effective means for the prevention of cervical cancer, widespread implementation of vaccination has been extremely difficult. Several potential issues have limited the development of widespread HPV vaccination programs, including cultural and religious beliefs, and limitations in the practicality of administering the vaccine. The overall goals of our work are to improve access to preventive strategies for cervical cancer. In this proposal we will examine the strategy of HPV vaccination for women who have just given birth. We believe that HPV vaccination of these women will be associated with a high level of patient satisfaction and acceptance. If successful, this strategy could play a major role in advancing the acceptance and implementation of HPV vaccination in the United States.

DETAILED DESCRIPTION:
Primary Objective

1. To estimate compliance with the HPV vaccine series when initiated in postpartum women.

Secondary Objectives

1. To determine patient acceptance and satisfaction with HPV vaccination administered in the postpartum period.
2. To determine predictors of compliance with the HPV vaccination series.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-26 years.
* Patients hospitalized during the postpartum period after a normal spontaneous vaginal delivery, assisted vaginal delivery or Cesarean section.
* Patients who delivered a singleton fetus or multiple gestations are eligible for participation.
* Patients may have delivered at gestational ages 32-44 weeks.
* Patients must have signed informed consent.
* Patients must meet pre-entry criteria.
* Patients who are breast feeding are eligible for participation.
* Patients must have an obstetrician whom they have seen for obstetric care and plan to follow-up with in the postpartum period.

Exclusion Criteria:

* Age < 18 or > 26 years.
* Patients with hemophilia, other bleeding disorders or thrombocytopenia (platelets < 100,000/ul).
* Patients receiving active anticoagulant therapy with warfarin, heparin or low molecular weight heparin.
* Pregnancy or planning pregnancy within the next 6 months.
* Ongoing bacteremia, endomyometritis or other serious febrile illness.
* Hypersensitivity to yeast, aluminum or other vaccine components.
* Prior vaccination with a prophylactic HPV vaccine (single or multiple doses).
* Patients who delivered a non-viable infant or an infant with severe congenital malformations.
* Patients who do not plan on following up postpartum with their local obstetrician or maternal fetal medicine specialist.
* Patients who are unwilling to receive subsequent doses of the HPV vaccine.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women, aged 18-26, hospitalized during the postpartum period after a normal spontaneous vaginal delivery, assisted vaginal delivery or Cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wright, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Walboomers JM, Jacobs MV, Manos MM, Bosch FX, Kummer JA, Shah KV, Snijders PJ, Peto J, Meijer CJ, Munoz N. Human papillomavirus is a necessary cause of invasive cervical cancer worldwide. J Pathol. 1999 Sep;189(1):12-9. doi: 10.1002/(SICI)1096-9896(199909)189:13.0.CO;2-F. PMID 10451482
- [Background] Schiffman M, Castle PE, Jeronimo J, Rodriguez AC, Wacholder S. Human papillomavirus and cervical cancer. Lancet. 2007 Sep 8;370(9590):890-907. doi: 10.1016/S0140-6736(07)61416-0. PMID 17826171
- [Background] FUTURE II Study Group. Quadrivalent vaccine against human papillomavirus to prevent high-grade cervical lesions. N Engl J Med. 2007 May 10;356(19):1915-27. doi: 10.1056/NEJMoa061741. PMID 17494925
- [Background] Garland SM, Hernandez-Avila M, Wheeler CM, Perez G, Harper DM, Leodolter S, Tang GW, Ferris DG, Steben M, Bryan J, Taddeo FJ, Railkar R, Esser MT, Sings HL, Nelson M, Boslego J, Sattler C, Barr E, Koutsky LA; Females United to Unilaterally Reduce Endo/Ectocervical Disease (FUTURE) I Investigators. Quadrivalent vaccine against human papillomavirus to prevent anogenital diseases. N Engl J Med. 2007 May 10;356(19):1928-43. doi: 10.1056/NEJMoa061760. PMID 17494926
- [Background] Joura EA, Leodolter S, Hernandez-Avila M, Wheeler CM, Perez G, Koutsky LA, Garland SM, Harper DM, Tang GW, Ferris DG, Steben M, Jones RW, Bryan J, Taddeo FJ, Bautista OM, Esser MT, Sings HL, Nelson M, Boslego JW, Sattler C, Barr E, Paavonen J. Efficacy of a quadrivalent prophylactic human papillomavirus (types 6, 11, 16, and 18) L1 virus-like-particle vaccine against high-grade vulval and vaginal lesions: a combined analysis of three randomised clinical trials. Lancet. 2007 May 19;369(9574):1693-702. doi: 10.1016/S0140-6736(07)60777-6. PMID 17512854
- [Background] Villa LL, Costa RL, Petta CA, Andrade RP, Ault KA, Giuliano AR, Wheeler CM, Koutsky LA, Malm C, Lehtinen M, Skjeldestad FE, Olsson SE, Steinwall M, Brown DR, Kurman RJ, Ronnett BM, Stoler MH, Ferenczy A, Harper DM, Tamms GM, Yu J, Lupinacci L, Railkar R, Taddeo FJ, Jansen KU, Esser MT, Sings HL, Saah AJ, Barr E. Prophylactic quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in young women: a randomised double-blind placebo-controlled multicentre phase II efficacy trial. Lancet Oncol. 2005 May;6(5):271-8. doi: 10.1016/S1470-2045(05)70101-7. PMID 15863374
- [Background] Koutsky LA, Ault KA, Wheeler CM, Brown DR, Barr E, Alvarez FB, Chiacchierini LM, Jansen KU; Proof of Principle Study Investigators. A controlled trial of a human papillomavirus type 16 vaccine. N Engl J Med. 2002 Nov 21;347(21):1645-51. doi: 10.1056/NEJMoa020586. PMID 12444178
- [Background] Markowitz LE, Dunne EF, Saraiya M, Lawson HW, Chesson H, Unger ER; Centers for Disease Control and Prevention (CDC); Advisory Committee on Immunization Practices (ACIP). Quadrivalent Human Papillomavirus Vaccine: Recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2007 Mar 23;56(RR-2):1-24. PMID 17380109
- [Background] Davis K, Dickman ED, Ferris D, Dias JK. Human papillomavirus vaccine acceptability among parents of 10- to 15-year-old adolescents. J Low Genit Tract Dis. 2004 Jul;8(3):188-94. doi: 10.1097/00128360-200407000-00005. PMID 15874862
- [Background] Lazcano-Ponce E, Rivera L, Arillo-Santillan E, Salmeron J, Hernandez-Avila M, Munoz N. Acceptability of a human papillomavirus (HPV) trial vaccine among mothers of adolescents in Cuernavaca, Mexico. Arch Med Res. 2001 May-Jun;32(3):243-7. doi: 10.1016/s0188-4409(01)00277-6. PMID 11395192
- [Background] Slomovitz BM, Sun CC, Frumovitz M, Soliman PT, Schmeler KM, Pearson HC, Berenson A, Ramirez PT, Lu KH, Bodurka DC. Are women ready for the HPV vaccine? Gynecol Oncol. 2006 Oct;103(1):151-4. doi: 10.1016/j.ygyno.2006.02.003. Epub 2006 Mar 21. PMID 16551476
- [Background] Taylor JA, Darden PM, Brooks DA, Hendricks JW, Wasserman RC, Bocian AB; Pediatric Research in Office Settings; National Medical Association. Association between parents' preferences and perceptions of barriers to vaccination and the immunization status of their children: a study from Pediatric Research in Office Settings and the National Medical Association. Pediatrics. 2002 Dec;110(6):1110-6. doi: 10.1542/peds.110.6.1110. PMID 12456907
- [Background] Tissot AM, Zimet GD, Rosenthal SL, Bernstein DI, Wetzel C, Kahn JA. Effective strategies for HPV vaccine delivery: the views of pediatricians. J Adolesc Health. 2007 Aug;41(2):119-25. doi: 10.1016/j.jadohealth.2007.05.007. PMID 17659214
- [Background] Kahn JA, Zimet GD, Bernstein DI, Riedesel JM, Lan D, Huang B, Rosenthal SL. Pediatricians' intention to administer human papillomavirus vaccine: the role of practice characteristics, knowledge, and attitudes. J Adolesc Health. 2005 Dec;37(6):502-10. doi: 10.1016/j.jadohealth.2005.07.014. PMID 16310128
- [Background] Daley MF, Liddon N, Crane LA, Beaty BL, Barrow J, Babbel C, Markowitz LE, Dunne EF, Stokley S, Dickinson LM, Berman S, Kempe A. A national survey of pediatrician knowledge and attitudes regarding human papillomavirus vaccination. Pediatrics. 2006 Dec;118(6):2280-9. doi: 10.1542/peds.2006-1946. PMID 17142510
- See also: Columbia University Department of Obstetrics and Gynecology — http://cumc.columbia.edu/dept/obgyn/gynonc/gynonc_team.html